CLINICAL TRIAL: NCT06336421
Title: The Effect of Virtual Reality Application on Perceived Anxiety and Vital Signs in Primiparous During Cesarean Section
Brief Title: The Effect of Virtual Reality Application on Perceived Anxiety and Vital Signs in Primiparous
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Ayse Aydin, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Şuletuvanç
Record Dates: First submitted 2024-03-22; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Cesarean Section Complications
Keywords: Virtual Reality; Cesarean; Primiparous; Anxiety; Vital Signs
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistics expert
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): virtual reality glasses were used in primiparous pregnant women undergoing cesarean section. The video, in which baby pictures will be shown accompanied by virtual reality music, was prepared by the researcher and a faculty member in the music department. During the cesarean section, the researcher showed the pregnant woman in the experimental group a video accompanied by music and baby pictures using virtual reality glasses for an average of 10 minutes.
  Interventions: Other: Virtual Reality
- Control group (No Intervention): * Written consent was obtained from pregnant women who agreed to participate in the study.
  * 10 minutes before cesarean section; A personal information form was filled out to determine the descriptive characteristics of the pregnant women.
  * The pregnant woman's anxiety level before the procedure was determined using the State Anxiety Scale.
  * Before the procedure, blood pressure, pulse, respiratory rate and saturation in the patient follow-up form were recorded.
  * Routine practice was performed during cesarean section.
  * 10 minutes after cesarean section; In order to determine the anxiety level, the parameters in the State Anxiety Scale and the Patient Follow-up Form were measured again and the process was completed.

INTERVENTIONS:
Other: Virtual Reality — VR Box brand virtual reality glasses were used in primiparous pregnant women undergoing cesarean section.
  During the cesarean section, the researcher showed the pregnant woman in the experimental group a video accompanied by music and baby pictures using virtual reality glasses for an average of 10 minutes.
  Arms: Experimental Group

SUMMARY:
Purpose: To determine the effect of virtual reality application on anxiety and vital signs perceived by primiparous women during cesarean section.The research was conducted in a randomized controlled experimental design.The population of the research consisted of primiparous pregnant women with a caesarean section indication in the Ataturk University Health Research and Application Center Gynecology Clinic Operating Room.

DETAILED DESCRIPTION:
Priority power analysis was performed to determine the size of the study. Cohen's standard field dimensions reference collection method was chosen in the image analysis. Medium effect size (0.5), alpha value compared to the base was determined as 5%, theoretical power was determined as 95% and the minimum volume was determined as 45. 90 pregnant women, 45 of whom were experimental and 45 of whom were controls, met the research criteria and did not agree to participate.Pregnant women in the sample were randomly assigned to two groups using random assignment by assigning them in numerical order.

Criteria for inclusion in the study;

* Having undergone epidural anesthesia, spinal anesthesia, combined anesthesia,
* Not having an emergency cesarean section,
* Being over 18 years of age,
* Being at least a primary school graduate,
* Not having been diagnosed with a high-risk pregnancy,
* Agreeing to participate in the research voluntarily,
* Not having any hearing or vision problems (for the experimental group),
* Not taking medications that affect blood pressure and pulse rate (such as digoxin, adrenaline, dopamine),
* No diagnosed psychiatric disease,
* Being primiparous,
* Being between 38-40 weeks of pregnancy. Exclusion criteria;
* Leaving the study at any stage of the research
* Patients who need general anesthesia during surgery. Pregnant women in the sample were randomly assigned to two groups using random assignment by giving them a numerical order. Then, it was decided by lottery method which group would be the experiment and which group would be the control. Since the data was collected by the researcher during the conduct of the study, blinding was not possible. However, while performing statistical analysis, nicknames were given to the experimental and control groups. Statistical analysis of the data was performed by an independent statistician blinded to the groups. After the analysis, interpretations were made by changing the group names. In this way, statistical bias was prevented during the data analysis step. Therefore, a single blinding technique was used. CONSORT 2010 Flow Diagram guidelines were followed during the research process."Personal Information Form", "State Anxiety Scale" and "Patient Follow-Up Form" were used to collect data in the study. Virtual reality was used as an intervention tool in the research.

ntervention Tool Used in the Research: Virtual Reality VR Box brand virtual reality glasses were used in primiparous pregnant women undergoing cesarean section. The video, in which baby pictures will be shown accompanied by virtual reality music, was prepared by the researcher and a faculty member in the music department. During the cesarean section, the researcher showed the pregnant woman in the experimental group a video accompanied by music and baby pictures using virtual reality glasses for an average of 10 minutes.

Data; It was collected face to face by the researcher at the Atatürk University Health Research and Application Center Obstetrics Clinic Operating Room between 01.11.2022 and 15.06.2023. It took an average of 5-10 minutes to fill out the forms.

Process steps Experimental group

* Written consent was obtained from pregnant women who agreed to participate in the study.
* 10 minutes before caesarean section; A personal information form was filled out to determine the descriptive characteristics of the pregnant women.
* Before cesarean section, anxiety level was determined with the State Anxiety Scale.
* Blood pressure, pulse, respiratory rate and saturation in the patient follow-up form were recorded.
* During the cesarean section, the pregnant woman was shown a video accompanied by music and baby pictures using virtual reality glasses for an average of 10 minutes.
* 10 minutes after cesarean section; In order to determine the anxiety level, the parameters in the State Anxiety Scale and the Patient Follow-up Form were measured again and the process was completed.

control group

* Written consent was obtained from pregnant women who agreed to participate in the study.
* 10 minutes before cesarean section; A personal information form was filled out to determine the descriptive characteristics of the pregnant women.
* The pregnant woman's anxiety level before the procedure was determined using the State Anxiety Scale.
* Before the procedure, blood pressure, pulse, respiratory rate and saturation in the patient follow-up form were recorded.
* Routine practice was performed during cesarean section.
* 10 minutes after cesarean section; In order to determine the anxiety level, the parameters in the State Anxiety Scale and the Patient Follow-up Form were measured again and the process was completed.

After data collection, evaluation and analysis were done in the SPSS 22 package statistics program. Normality distributions of the data were examined. Skewness-kurtosis values were examined to check whether the data conformed to normal distribution and it was determined that the values of all data were between -1.5 and +1.5. It was determined that parametric testing techniques could be applied. In the analysis of data; number, percentage distribution, mean, standard deviation, chi-square, Independent-samples t test and paired-samples t test were used.

ELIGIBILITY:
Inclusion Criteria:

* • Having undergone epidural anesthesia, spinal anesthesia, combined anesthesia,

  * Not having an emergency cesarean section,
  * Being over 18 years of age,
  * Being at least a primary school graduate,
  * Not having been diagnosed with a high-risk pregnancy,
  * Agreeing to participate in the research voluntarily,
  * Not having any hearing or vision problems (for the experimental group),
  * Not taking medications that affect blood pressure and pulse rate (such as digoxin, adrenaline, dopamine),
  * No diagnosed psychiatric disease,
  * Being primiparous,
  * Being between 38-40 weeks of pregnancy.

Exclusion Criteria:

* • Leaving the study at any stage of the research

  * Patients who need general anesthesia during surgery.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 90 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | 8 months
  There are 18 questions in this form, prepared by the researchers in line with the literature.
State Anxiety Scale | 8 months
  This scale was developed by Spielberger et al. Developed by. The adaptation of the scale to Turkish and its validity and reliability studies were carried out by Öner and Le Compte in 1983.The scale is a 4-point Likert scale consisting of the options "not at all", "somewhat", "a lot", "completely". There are 10 direct and 10 reversed statements in the scale. Positive (increasing the total anxiety score) for items 3, 4, 6, 7, 9, 12, 13, 14, 17, 18 in the scale; 1, 2, 5, 8, 10, 11, 15, 16, 19 Negative scores (reducing the total anxiety score) are obtained for the 20th items. The highest score is 80 and the lowest score is 20. A high total score indicates that the person's anxiety level is also high.Cronbach's alpha coefficient was found to be 0.79 for state anxiety. In this study, Cronbach's Alpha value was found to be 0.83.
Pregnant follow-up form | 8 months
  Blood pressure, pulse, respiration and the amount of oxygen in the blood were measured before and after the procedure and recorded on this form.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Aydın, Study Director — Ataturk University
Locations (1):
- Ayse Aydin, Yakutiye, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No